CLINICAL TRIAL: NCT00847561
Title: Family-Based Prevention for Childhood Anxiety
Brief Title: Effectiveness of a Family-Based Treatment for Preventing Anxiety Disorders in At-Risk Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Golda S. Ginsburg, Ph.D., Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH077312 (NIH); R01MH077312 (NIH); R01MH077312-01 (NIH); DDTR B4-TBI (Other: ClinicalTrials.gov)
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Anxiety Disorders
Keywords: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family-based CBT (Experimental): Family-based CBT. Participants will receive family-based cognitive behavioral therapy. Families in this group will learn about how to identify the signs and symptoms of anxiety, ways to cope with anxiety, relaxation techniques, and problem-solving skills. They will participate in 8, one-hour sessions, once/week with trained clinicians and 3 monthly booster sessions to reinforce what they learned.
  Interventions: Behavioral: Family-based CBT
- Information Monitoring (Placebo Comparator): Information Monitoring. Participants will receive a packet of information about anxiety. Participants in this group will be called monthly to monitor symptoms of anxiety.
  Interventions: Behavioral: Information Monitoring

INTERVENTIONS:
Behavioral: Family-based CBT — Eight, 1-hour weekly sessions with a trained clinician.
  Arms: Family-based CBT
Behavioral: Information Monitoring — Packet providing information on strategies for coping with anxiety
  Arms: Information Monitoring

SUMMARY:
This study will test the effectiveness of a family-based, cognitive behavioral therapy (CBT)-based program for preventing anxiety disorders in at-risk children.

DETAILED DESCRIPTION:
Anxiety disorders are among the most common mental disorders in children and adolescents, and they are associated with short- and long-term impairment in social, academic, familial, and psychological functioning. The children of parents with anxiety disorders are more likely to develop anxiety disorders themselves, because of genetic factors and the atmosphere in which they are raised. Previous research indicates that the risk of anxiety disorders among children can be reduced through preventive therapeutic interventions. In children with anxiety disorders whose parents also have anxiety disorders, therapy that includes their family is more successful than therapy focused only on the child. This study will test the effectiveness of a preventive, family-based therapy for children whose parents have anxiety disorders.

Participation in this study will last 1 year. First, interested participants will be asked to perform a screening assessment. This will include providing information about the symptoms, behaviors, and functioning of parent and child participants; filling out questionnaires; and videotaping the child and parent participants interacting. If, after the screening, participants are selected to continue with the study, they will be randomly assigned to receive either information monitoring or family-based cognitive behavioral therapy. Child and parent participants assigned to information monitoring will receive a booklet with information on coping with anxiety. Child and parent participants assigned to family-based cognitive behavioral therapy will meet with a study clinician for eight, weekly, 1-hour intervention visits, during which participants will learn skills to reduce anxiety. After completing the weekly visits, participants in this group will also receive three monthly booster sessions, in which coping skills will be reviewed. In addition to the screening visit, all participants will undergo identical assessments at three more time periods: 9 weeks, 6 months, and 12 months after entering the study. All participants will also receive monthly phone calls throughout the study to monitor the children's anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Parents of child participant have a current, primary anxiety disorder

Exclusion Criteria:

* Child has an anxiety disorder or is currently in treatment for anxiety

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2008-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Golda S. Ginsburg, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Slade EP, Ginsburg GS, Riddle MA. Cost-benefit Analysis of the Coping and Promoting Strength Program. Prev Sci. 2021 Nov;22(8):1096-1107. doi: 10.1007/s11121-021-01309-5. Epub 2021 Oct 14. PMID 34647197
- [Derived] Ginsburg GS, Tein JY, Riddle MA. Preventing the Onset of Anxiety Disorders in Offspring of Anxious Parents: A Six-Year Follow-up. Child Psychiatry Hum Dev. 2021 Aug;52(4):751-760. doi: 10.1007/s10578-020-01080-8. Epub 2020 Oct 18. PMID 33070244
- [Derived] Schleider JL, Ginsburg GS, Drake K. Perceived Peer Victimization Predicts Anxiety Outcomes in a Prevention Program for Offspring of Anxious Parents. J Clin Child Adolesc Psychol. 2018;47(sup1):S255-S263. doi: 10.1080/15374416.2016.1270831. Epub 2017 Feb 1. PMID 28145769
- [Derived] Ginsburg GS, Drake KL, Tein JY, Teetsel R, Riddle MA. Preventing Onset of Anxiety Disorders in Offspring of Anxious Parents: A Randomized Controlled Trial of a Family-Based Intervention. Am J Psychiatry. 2015 Dec;172(12):1207-14. doi: 10.1176/appi.ajp.2015.14091178. Epub 2015 Sep 25. PMID 26404420

RESULTS

PARTICIPANT FLOW:
Groups:
- Family-based CBT: Family-based Cognitive Behavioral Therapy (CBT). Participants will receive family-based cognitive behavioral therapy. Families in this group will learn about how to identify the signs and symptoms of anxiety, ways to cope with anxiety, relaxation techniques, and problem-solving skills. They will participate in 8, one-hour sessions, once/week with trained clinicians and 3 monthly booster sessions to reinforce what they learned.
  Family-based CBT: Eight, 1-hour weekly sessions with a trained clinician.
Period: Overall Study
Arm/Group | Family-based CBT | Information Monitoring
Started | 70 | 66
Completed | 57 | 62
Not Completed | 13 | 4
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Unable to schedule | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Family-based CBT | Information Monitoring | Total
Number analyzed (Participants) | 70 | 66 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.53 (7.76) | 8.86 (1.85) | 8.69 (1.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 32 | 76
  Male | 26 | 34 | 60
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 58 | 57 | 115
  other ethnicity/race | 12 | 9 | 21
Region of Enrollment [Number; unit: participants]
  United States | 70 | 66 | 136

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Disorders Interview Schedule for Diagnostic and Statistical Manual for Psychological Disorders-IV, Child and Parent Versions (C/P-ADIS)
Description: The C/P-ADIS is a semi-structured diagnostic interview used to assess symptoms of anxiety, depression, and behavioral issues.
  This interview will be administered by a trained staff member and will utilize information from both parents and children.
  This interview will be used to determine the presence or absence of an anxiety disorder for children in this study.
  .
Time Frame: 12 months post-treatment
Measure: Number; unit: participants with anxiety diagnosis
Arm/Group | Information Monitoring | Family-based CBT
Number analyzed (Participants) | 66 | 70
participants with anxiety diagnosis | 19 | 3

ADVERSE EVENTS:
Arm/Group | Family-based CBT | Information Monitoring
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/66
Other Adverse Events (participants affected / at risk) | 0/70 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes